CLINICAL TRIAL: NCT02715258
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Compare the Efficacy and Safety of Bexagliflozin to Placebo in Subjects With Type 2 Diabetes Mellitus and Inadequate Glycemic Control
Brief Title: Safety and Efficacy of Bexagliflozin as Monotherapy in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THR-1442-C-450
Record Dates: First submitted 2016-03-11; First posted 2016-03-22 (Estimated); Results first posted 2021-04-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — bexagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bexagliflozin tablets, 20 mg (Active Comparator): Each subject will self-administer bexagliflozin tablets once daily for 24 weeks.
  Interventions: Drug: Bexagliflozin
- Placebo tablets (Placebo Comparator): Each subject will self-administer placebo (inactive tablet) once daily for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bexagliflozin — tablets containing 20 mg bexagliflozin
  Other Names: EGT0001442
  Arms: Bexagliflozin tablets, 20 mg
Drug: Placebo — tablets matching the appearance of bexagliflozin tablets
  Arms: Placebo tablets

SUMMARY:
The purpose of this study is to investigate the effect of bexagliflozin in lowering hemoglobin A1c (HbA1c) levels in patients with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This was a phase 3, multi-center, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of once daily oral administration of bexagliflozin tablets, 20 mg or placebo tablets, in male and female subjects with T2DM who were treatment-naïve or previously treated with 1 oral hypoglycemic agent (OHA).

Prospective subjects being treated with one OHA were eligible if they had an HbA1c between 6.5% and 10.0% and were willing to complete a 6-week washout. Individuals taking thiazolidinediones were not eligible for the study. All eligible subjects were to start a 2-week placebo run-in period. Subjects who missed no more than 1 dose of the run-in medication, had fasting blood glucose values ≥ 250 mg/dL on no more than two consecutive days, and had an HbA1c level between 7.0% and 10.5% and a fasting glucose level < 250 mg/dL after the run-in period were eligible for randomization.

Two hundred and ten (210) subjects were planned to be randomly assigned to receive oral bexagliflozin tablets, 20 mg or placebo, in a 2:1 ratio once daily for 24 weeks. Subjects with uncontrolled hyperglycemia based on blood glucose levels could receive additional approved anti-diabetic medications. Treatment group assignment at the start of the treatment period was stratified by baseline HbA1c level and background anti-diabetes treatment status (treatment naïve or not).

Each subject was contacted by telephone at week 2 and was instructed to return to the clinic at weeks 6, 12, 18, and 24 for efficacy assessment and safety monitoring. Subjects returned to the clinic for a follow-up visit at week 26 or 2 weeks after the last dose of investigational product if the subject terminated prior to week 24.

ELIGIBILITY:
The study population included:

1. Male or female adult subjects ≥ 18 years of age at screening
2. Subjects who were treatment naïve or receiving 1 OHA in combination with diet and exercise
3. Subjects with a diagnosis of T2DM
4. Subjects with HbA1c levels at screening between 7.0% and 10.5% (inclusive) if treatment-naïve or with HbA1c levels between 6.5 and 10.0% (inclusive) if on 1 oral anti diabetic agent
5. Subjects with a BMI ≤ 45 kg/m2
6. Subjects whose doses of medications for hypertension or hyperlipidemia (if applicable) had not changed for at least 30 days prior to screening
7. Subjects who were willing and able to return for all clinic visits and to complete all study required procedures
8. Female subjects of childbearing potential who were willing to use an adequate method of contraception and not become pregnant for the duration of the study.
9. Subjects who maintained glycemic control throughout washout, if applicable.
10. Subjects who had HbA1c levels between 7.0 and 10.5% prior to randomization
11. Subjects who had been compliant in investigational product administration by missing no more than 1 dose of run-in medication

Subjects who met any of the following criteria were excluded from the study:

1. A diagnosis of type 1 diabetes mellitus or maturity-onset diabetes of the young
2. Use of injected therapy for treatment of diabetes (insulin or GLP-1 receptor agonist therapy) or thiazolidinedione class drugs at the time of screening
3. Female subjects who were pregnant or breastfeeding
4. Hemoglobinopathy or carrier status for hemoglobin alleles that affected HbA1c measurement
5. Genitourinary tract infection (e.g., UTI, GMI, vaginitis, balanitis) within 6 weeks of screening or history of ≥ 3 genitourinary infections requiring treatment within 6 months from screening
6. Estimated glomerular filtration rate (eGFR), as calculated by the modification of diet in renal disease study equation (MDRD), < 60 mL/min/1.73 m2 at screening
7. Uncontrolled hypertension defined as a sitting systolic blood pressure >160 mm Hg or diastolic blood pressure > 95 mm Hg at screening
8. A positive result for hepatitis B surface antigen (HBsAg) or hepatitis C (HCV)
9. History of alcohol or illicit drug abuse in the past 2 years
10. Known human immunodeficiency virus (HIV) positive based on medical history
11. Life expectancy < 2 years
12. New York Heart Association (NYHA) Class IV heart failure within 3 months of screening
13. MI, unstable angina, stroke, or hospitalization for heart failure within 3 months of screening
14. Treatment with an investigational drug within 30 days or within 7 half-lives of the investigational drug, whichever was longer
15. Previous treatment with bexagliflozin or EGT0001474
16. Use of any SGLT2 inhibitors, either at the time of screening or in the prior 3 months
17. Currently participating in another interventional trial
18. Not able to comply with the study scheduled visits
19. Any condition, disease, disorder, or clinically relevant abnormality that, in the opinion of the primary investigator, would jeopardize the subject's appropriate participation in this study or obscure the effects of treatment
20. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 x ULN or total bilirubin ≥ 1.5 x upper limit of normal (ULN) with the exception of isolated Gilbert's syndrome at screening
21. Two or more consecutive FPG measures ≥ 250 mg/dL (13.9 mmol/L) prior to randomization or severe clinical signs or symptoms of hyperglycemia during the washout or run-in periods, including weight loss, blurred vision, increased thirst, or increased urination, or fatigue
22. At last visit prior to randomization, FPG level ≥ 250 mg/dL
23. Prior renal transplantation or evidence of nephrotic syndrome (defined as a urine albumin-to-creatinine ratio (UACR) > 2000 mg/g at screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Paul Lock, MD, Study Director — Theracos
Locations (23):
- United States (18):
  - Research Site, Canoga Park, California
  - Research Site, Chino, California
  - Research Site, Huntington Park, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Orlando, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Trenton, New Jersey
  - Research Site, Calabash, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Munroe Falls, Ohio
  - Research Site, Portland, Oregon
  - Research Site, North Myrtle Beach, South Carolina
  - Research Site, DeSoto, Texas
  - Research Site, Fort Worth, Texas
- Canada (5):
  - Research Site, Vancouver, British Columbia
  - Research Site, Newmarket, Ontario
  - Research Site 2, Toronto, Ontario
  - Research Site 1, Toronto, Ontario
  - Research Site, Pointe-Claire, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 210 subjects were randomized to be in the bexagliflozin arm or in the placebo arm in a ratio of 2:1.
Groups:
- Bexagliflozin Tablets, 20 mg: Each subject will receive bexagliflozin tablets, 20 mg once daily for 24 weeks.
- Placebo Tablets: Each subject will receive placebo (inactive tablet) once daily for 24 weeks.
Period: Overall Study
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Started | 140 | 70
Intent to Treat/Safety Analysis (Three randomized subject numbers were excluded in the ITT and the safety populations due to GCP violation.) | 138 | 69
Completed | 124 | 64
Not Completed | 16 | 6
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Lost to Follow-up | 7 | 1
Not completed — Terminated by Sponsor | 0 | 1
Not completed — Death | 0 | 1
Not completed — Subject non-compliant | 1 | 1
Not completed — GCP violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets | Total
Number analyzed (Participants) | 138 | 69 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (10.21) | 54.7 (11.02) | 55.4 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 35 | 107
  Male | 66 | 34 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67 | 40 | 107
  Not Hispanic or Latino | 71 | 29 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 5 | 20
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 25 | 6 | 31
  White | 96 | 58 | 154
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 21 | 12 | 33
  United States | 117 | 57 | 174
Body Weight at Baseline [Mean (Standard Deviation); unit: kg] | 90.5 (20.48) | 84.6 (19.75) | 88.6 (20.39)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.79 (5.653) | 30.48 (4.650) | 32.01 (5.437)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 131.0 (14.35) | 125.6 (13.84) | 129.2 (14.38)
HbA1c [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 8.05 (0.824) | 7.97 (0.757) | 8.02 (0.801)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.39 (1.957) | 9.45 (2.079) | 9.41 (1.994)
Duration of Diabetes from Diagnosis to Screening [Mean (Standard Deviation); unit: years] | 5.9 (5.82) | 6.5 (5.21) | 6.1 (5.62)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline at Week 24
Description: Glycated hemoglobin A1c (%) was measured using an HPLC method in the laboratories that had completed NGSP Level I laboratory certification and were traceable to the Diabetes Control and Complications Trial (DCCT) reference method.
Time Frame: 24 weeks
Population: Intention-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: % of HbA1c
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 138 | 69
% of HbA1c | -0.51 (0.082) | -0.10 (0.108)
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Analysis of change from baseline in HbA1c (%) at Week 24; Test type: Superiority; p = 0.0012, Mixed Models Analysis — The mixed-effects repeated measures analysis includes country, background anti-diabetes treatment status, treatment, visit, treatment-by-visit interaction and the baseline HbA1c value as a fixed effect covariate; mixed-effects repeated measures = -0.41, 95% CI 2-sided [-0.66 to -0.16]
Statistical Analysis 2: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Sensitivity Analysis 1: Multiple imputation for change from baseline in HbA1c (%) including observations obtained after rescue medication; Test type: Superiority; p = 0.0021, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -0.41, 95% CI 2-sided [-0.68 to -0.15]
Statistical Analysis 3: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Sensitivity Analysis 2: Multiple imputation for change from baseline in HbA1c (%) excluding observations obtained after rescue medication; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -0.55, 95% CI 2-sided [-0.80 to -0.30]
Statistical Analysis 4: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Sensitivity Analysis 3: LOCF for change from baseline in HbA1c (%) including observations obtained after rescue medication; Test type: Superiority; p = 0.0009, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -0.40, 95% CI 2-sided [-0.64 to -0.17]

2. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline at Week 24
Description: Blood pressure (BP) measurements are obtained using a calibrated sphygmomanometer in sitting, supine and standing positions. The left arm and same cuff sizes should be used for each measurement at all visits. If the left arm cannot be used at the screening visit or during the study for BP measurements, the reason should be documented and the right arm should be used for BP measurements for all subsequent visits.
Time Frame: 24 weeks
Population: ITT analysis set
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 138 | 69
mmHg | -0.60 (1.145) | 1.54 (1.524)
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Analysis of change from baseline in SBP (mm Hg) at Week 24; Test type: Superiority; p = 0.2340, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -2.14, 95% CI 2-sided [-5.66 to 1.39]
Statistical Analysis 2: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Sensitivity Analysis 1: Multiple imputation for change from baseline in SBP (mm Hg) including observations obtained after rescue medication; Test type: Superiority; p = 0.2937, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -1.91, 95% CI 2-sided [-5.48 to 1.66]
Statistical Analysis 3: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Sensitivity Analysis 2: Multiple imputation for change from baseline in SBP (mm Hg) excluding observations obtained after rescue medication; Test type: Superiority; p = 0.4030, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -1.72, 95% CI 2-sided [-5.75 to 2.32]
Statistical Analysis 4: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.2160, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -2.09, 95% CI 2-sided [-5.41 to 1.23]

3. Secondary Outcome: Change in Body Weight From Baseline at Week 24 in Subjects With a BMI ≥ 25 Kg/m2
Description: The body weight was obtained using a calibrated scale as part of complete physical examination or abbreviated physical examination.
Time Frame: 24 weeks
Population: Subjects with BMI >= 25 kg/m2 in the ITT analysis set
Measure: Least Squares Mean (Standard Error); unit: Kg
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 128 | 62
Kg | -1.85 (0.394) | -1.06 (0.485)
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Analysis of change from baseline in body weight (kg) at Week 24 for subjects with BMI greater than or equal to 25 kg/m2; Test type: Superiority; p = 0.1222, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -0.79, 95% CI 2-sided [-1.80 to 0.21]
Statistical Analysis 2: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Sensitivity Analysis 1: Multiple imputation for change from baseline in body weight (kg) for subjects with BMI greater than or equal to 25 kg/m2 including observations obtained after rescue medication; Test type: Superiority; p = 0.2014, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -0.65, 95% CI 2-sided [-1.65 to 0.35]
Statistical Analysis 3: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Sensitivity Analysis 2: Multiple imputation for change from baseline in body weight (kg) for subjects with BMI greater than or equal to 25 kg/m2 excluding observations obtained after rescue medication; Test type: Superiority; p = 0.0638, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -0.91, 95% CI 2-sided [-1.88 to 0.05]
Statistical Analysis 4: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Sensitivity Analysis 3: LOCF for change from baseline in body weight (kg) for subjects with BMI greater than or equal to 25 kg/m2 including observations obtained after rescue medication; Test type: Superiority; p = 0.1456, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -0.69, 95% CI 2-sided [-1.63 to 0.24]

4. Other Pre Specified Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) Over Time
Description: The fasting plasma glucose (FPG) is measured at each study visit. The subject must have fasted for approximately 10 hours prior to the blood draw to ensure that the FPG value is truly a fasting sample.
Time Frame: 24 weeks
Population: Subjects with a value at baseline and Week 6, 12, 18 and 24
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 133 | 65
mmol/L
  Change from baseline at Week 6 | -1.40 (2.116) | 0.50 (2.655)
  Change from baseline at Week 12: number analyzed (Participants) | 132 | 64
  Change from baseline at Week 12 | -1.41 (1.904) | 0.33 (2.103)
  Change from baseline at Week 18: number analyzed (Participants) | 127 | 63
  Change from baseline at Week 18 | -1.17 (2.058) | 0.03 (2.337)
  Change from baseline at Week 24: number analyzed (Participants) | 125 | 64
  Change from baseline at Week 24 | -1.02 (2.013) | -0.15 (2.480)
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Analysis of change from baseline in FPG (mmol/L) over time across 24 weeks; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -1.50, 95% CI 2-sided [-1.92 to -1.09]

5. Other Pre Specified Outcome: Change From Baseline of HbA1c From Baseline Over Time
Description: as for outcome 1
Time Frame: 24 weeks
Population: Subjects with a value at baseline and at Week 6, 12, 18 and 24
Measure: Least Squares Mean (Standard Error); unit: % of HbA1c
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 133 | 65
% of HbA1c
  Change from baseline at Week 6 | -0.47 (0.064) | 0.13 (0.082)
  Change from baseline at Week 12: number analyzed (Participants) | 131 | 64
  Change from baseline at Week 12 | -0.61 (0.072) | 0.10 (0.095)
  Change from baseline at Week 18: number analyzed (Participants) | 127 | 63
  Change from baseline at Week 18 | -0.58 (0.071) | -0.01 (0.093)
  Change from baseline at Week 24 | -0.51 (0.082) | -0.10 (0.108)
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Change from baseline in HbA1c (%) at Week 6; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -0.61, 95% CI 2-sided [-0.79 to -0.43]
Statistical Analysis 2: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Change from baseline in HbA1c (%) at Week 12; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -0.71, 95% CI 2-sided [-0.92 to -0.50]
Statistical Analysis 3: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Change from baseline in HbA1c (%) at Week 18; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -0.57, 95% CI 2-sided [-0.78 to -0.36]
Statistical Analysis 4: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Change from baseline in HbA1c (%) at Week 24; Test type: Superiority; p = 0.0012, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -0.41, 95% CI 2-sided [-0.66 to -0.16]
Statistical Analysis 5: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Change from baseline in HbA1c (%) across 24 weeks; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; mixed-effects repeated measures = -0.58, 95% CI 2-sided [-0.76 to -0.39]

6. Other Pre Specified Outcome: Proportion of Subjects Who Achieve an HbA1c < 7%
Description: as for outcome 1
Time Frame: Up to 24 weeks
Population: Subjects with a value at baseline and at Week 6, 12, 18 and 24
Measure: Number; unit: participants
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 133 | 65
participants
  Proportion of subjects with HbA1c < 7% at Week 6 | 35 | 6
  Proportion of subjects with HbA1c < 7% at Week 12: number analyzed (Participants) | 131 | 64
  Proportion of subjects with HbA1c < 7% at Week 12 | 44 | 8
  Proportion of subjects with HbA1c < 7% at Week 18: number analyzed (Participants) | 127 | 63
  Proportion of subjects with HbA1c < 7% at Week 18 | 42 | 10
  Proportion of subjects with HbA1c < 7% at Week 24: number analyzed (Participants) | 124 | 64
  Proportion of subjects with HbA1c < 7% at Week 24 | 41 | 13
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Model-Adjusted proportion of subjects with HbA1c <7% across 24 weeks; Test type: Superiority; p = 0.0006, ANCOVA — The logistic regression includes country, background anti-diabetes treatment status, treatment, visit, treatment-by-visit interaction and the baseline HbA1c value as a fixed effect covariate; Odds Ratio (OR) = 3.39, 95% CI 2-sided [1.69 to 6.80]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from -8 weeks (V2) to 26 weeks (V12) according to the Schedule of Events outlined in the study protocol. Subjects in the Bexagliflozin group had mean study drug exposure of 22.52 weeks and the placebo group had mean mean study drug exposure of 22.90 weeks.
Groups:
- Bexagliflozin Tablets, 20 mg: Each subject was to take bexagliflozin tablets, 20 mg once daily for 24 weeks.
- Placebo Tablets: Each subject was to take placebo (inactive tablet) once daily for 24 weeks.
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
All-Cause Mortality (participants affected / at risk) | 0/138 | 1/69
Serious Adverse Events (participants affected / at risk) | 1/138 | 1/69
Other Adverse Events (participants affected / at risk) | 41/138 | 25/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexagliflozin Tablets, 20 mg (N=138) | Placebo Tablets (N=69)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexagliflozin Tablets, 20 mg (N=138) | Placebo Tablets (N=69)
Urinary tract infection (Infections and infestations) | 7 (7) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Polyuria (Renal and urinary disorders) | 10 (10) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 4 (5) | 5 (5)
Fatigue (General disorders) | 5 (5) | 0 (0)
Hypertension (Vascular disorders) | 3 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator does not have the right to publish the results.

DOCUMENTS (2):
  • Study Protocol (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT02715258/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT02715258/SAP_001.pdf